CLINICAL TRIAL: NCT04408664
Title: WP3-Influence of Cromones on EVH-test in Young (Elite) Athletes Who Tested Positive for EIB (=Exercise Induced Bronchoconstriction)
Brief Title: Influence of Cromones on Eucapnic Hyperventilation (EVH)-Test in Young (Elite) Athletes Who Tested Positive for EIB.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Jessa Hospital (Other); Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: s63147
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Exercise-Induced Bronchoconstriction
Keywords: Athletes; Sodium Cromoglycate; Cromones; Lomudal
MeSH Terms: interventions — Cromolyn Sodium; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Cromoglycate (Experimental): Patients will take Sodium Cromoglycate (SCG) (Lomudal®) 4 times daily during 6 months: SCG 4X1 ampulla of 2 mL daily (by Omron pocket aerosol).
  Interventions: Drug: Sodium Cromoglycate
- Sodium Chloride 0.9% (Placebo Comparator): Patients will take Sodium Chloride 0.9% 4 times daily during 6 months: Sodium Chloride 4X1 ampulla of 2 mL daily (by Omron pocket aerosol).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Cromoglycate — Sodium Cromoglicate 10 mg/mL packed in ampulla of 2 mL; Daily dosis of 4X20 mg milligram delivered by aerosol.
  Other Names: DNCG Iso; Lomudal
  Arms: Sodium Cromoglycate
Drug: Placebo — Sodium Chloride 0.9% packed in ampulla of 2 mL; Daily dosis of 4 ampulla delivered by aerosol.
  Other Names: Sodium Chloride
  Arms: Sodium Chloride 0.9%

SUMMARY:
This is a randomized, double-blinded, placebo-controlled trial of nebulized Sodium Cromoglycate (SCG) (Lomudal®) versus NaCl0.9% in athletes (11-18 year) with exercise-induced bronchoconstriction (EIB).

DETAILED DESCRIPTION:
Screening and diagnosing EIB (studied by investigators in WP1 (s59778) and WP2 (s61602) of granted FWO-TBM project (T001417N)) in young athletes would only be useful if a safe and effective treatment is available. Sodium Cromoglycate (SCG) has a very nice safety profile but is less effective when compared to inhaled corticosteroids in asthma patients. However, SCG has been shown to be especially effective in exercise-induced asthma and to reduce metabolite secretion in athletes due to hyperpnoea. Although commercial interest in the drug has fainted, from a clinical point of view, it remains the ideal candidate to be used in adolescents with features of EIB at risk to develop asthma in whom today no treatment would be initiated.

This clinical trial (s63147), which is WP3 of the FWO-TBM project, is a randomized double-blinded trial with subjects who tested positive for the diagnosis of EIB in either WP1 or WP2. Subjects who gave assent and whose parents gave consent will be randomized (1/1) in a double-blinded trial to receive either (arm 1) Sodium Cromoglycate (SCG) (Lomudal®) or (arm 2) placebo, both 4X1 ampulla (2 mL) in aerosol daily, during 6 months.

During the previous trials, several tests were already performed. If subjects want to participate in this trial and the previous tests were more than 1 month ago, some tests will be repeated as a baseline: questionnaires, spirometry (with reversibility test) and EVH-test. After 3 months, regular intake as well as potential side effects will be evaluated. After 6 months, in addition to questionnaires, clinical examination and spirometry with reversibility test, the EVH-test will be repeated. Subjects will also be offered the possibility to repeat (as they did for WP1 and WP2) a blood and sputum sampling at 6 months. Afterwards, subjects will have the option to continue open-label treatment for 6 months.

The investigators want to investigate the influence of SCG on EVH-test in young athletes who tested positive for EIB.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of exercise-induced-bronchoconstriction (EIB) based on positive EVH-test in WP1 (s59778) or WP2 (s61602)
* BMI between 5th and <85th percentile for age and gender

Exclusion Criteria:

* Clinically diagnosed asthma
* Baseline lung function:

  * FEV1%: ≤80% predicted FEV1%
  * Tiffeneau: FEV1/FVC% < 85%
  * Salbutamol-induced FEV1 reversibility ≥ 12%
* Any disorder, which in the investigator's opinion might jeopardize participant's safety or compliance with the protocol
* Smoker
* Participation in other study related to IMP
* If applicable: female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change in percentage maximal fall of FEV1 after EVH-test compared to baseline maximal fall | 6 months
  Individual's paired change in percentage maximal fall of FEV1 in relation to EVH-test between baseline values and values after 6 month treatment with sodium cromoglycate or placebo.

SECONDARY OUTCOMES:
Difference in symptom perception on a scale 0 to 5, with 5 maximum score per symptom | 6 months
  Symptom perception will be assessed by a questionnaire (scale: no, very mild, little, moderate, serious, very serious) . Comparison will be done per individual and between both arms.
Asthma development | 6 months
  Asthma development will be assessed by the occurrence of a positive reversibility test during the trial and compared between both arms.
Biomarkers in blood/sputum (optional) | 6 months
  Change in expression of inflammatory markers and markers of epithelial damage after 6 months of treatment in blood and sputum (e.g. CC16, uric acid, IL1-B, ...)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Maria Middelares, Ghent

IPD SHARING:
Plan to Share IPD: No
data will be analysed and grouped before release

REFERENCES:
- [Background] Van der Eycken S, Schelpe A, Marijsse G, Dilissen E, Troosters T, Vanbelle V, Aertgeerts S, Dupont LJ, Peers K, Bullens DM, Seys SF. Feasibility to apply eucapnic voluntary hyperventilation in young elite athletes. Respir Med. 2016 Feb;111:91-3. doi: 10.1016/j.rmed.2015.12.012. Epub 2016 Jan 4. PMID 26790574
- [Background] Jonckheere AC, Seys S, Dilissen E, Schelpe AS, Van der Eycken S, Corthout S, Verhalle T, Goossens J, Vanbelle V, Aertgeerts S, Troosters T, Peers K, Dupont L, Bullens D. Early-onset airway damage in early-career elite athletes: A risk factor for exercise-induced bronchoconstriction. J Allergy Clin Immunol. 2019 Nov;144(5):1423-1425.e9. doi: 10.1016/j.jaci.2019.07.014. Epub 2019 Jul 26. No abstract available. PMID 31356920
- [Background] Kippelen P, Larsson J, Anderson SD, Brannan JD, Dahlen B, Dahlen SE. Effect of sodium cromoglycate on mast cell mediators during hyperpnea in athletes. Med Sci Sports Exerc. 2010 Oct;42(10):1853-60. doi: 10.1249/MSS.0b013e3181da4f7d. PMID 20216468